CLINICAL TRIAL: NCT04502433
Title: Multicenter, Open-label, Randomised Trial to Assess the Efficacy and Tolerability of Poractant Alfa(Porcine Surfactant, Curosurf®) in Hospitalized Patients With SARS-COV-19 Acute Respiratory Distress Syndrome (ARDS)
Brief Title: Poractant Alfa (Curosurf®)) -- Effect in Adult Patients Diagnosed With 2019 Novel Coronavirus (SARS-COV-19; (Covid-19)) Acute Respiratory Distress Syndrome (ARDS)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The enrolment was extended. Nevertheless, despite the Sponsor's attempts, the infection status did not permit the identification of eligible patients for the study to complete it in a reasonable time.
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLI-050000-04; 2020-002632-75 (EudraCT Number)
Record Dates: First submitted 2020-08-03; First posted 2020-08-06 (Actual); Results first posted 2023-06-23 (Actual); Last update posted 2023-06-23 (Actual); Status verified 2023-05

CONDITIONS: Acute Respiratory Distress Syndrome
Keywords: acute respiratory distress syndrome; ARDS; Adults; Surfactant; Poractant alfa (porcine surfactant, Curosurf®),; Curosurf®; Coronavirus disease (COVID-19); Coronavirus 2019 Disease
MeSH Terms: conditions — Respiratory Distress Syndrome; COVID-19 | interventions — poractant alfa

STUDY DESIGN:
Intervention Model Description: Seventy patients will be randomized in the study with a ratio 3:2 (i.e. 42 patients in the poractant alfa arm and 28 in the control arm).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Patients treated with standard-of-care (SoC), as control cohort
- Poractant alfa (Experimental): Patients treated with CUROSURF® (poractant alfa), as an add-on to standard-of-care (SoC)
  Interventions: Drug: CUROSURF® (poractant alfa)

INTERVENTIONS:
Drug: CUROSURF® (poractant alfa) — Three administrations with a 24 hours dosing interval.
  Each endotracheal (ET) administration 1, 2, and 3 consisted of poractant alfa bolus:
  30mg /kg (Lean Body Weight-LBW) = 0.375ml /kg LBW, diluted with normal saline up to 2ml /kg LBW.
  Arms: Poractant alfa

SUMMARY:
The purpose of this study was to evaluate the efficacy and safety of poractant alfa (Curosurf®), administered by endotracheal (ET) instillation in hospitalized adult patients diagnosed with SARS-COV-19 acute respiratory distress syndrome (ARDS).

DETAILED DESCRIPTION:
This was a multicentre, open-label, randomized phase II proof-of-concept study.

The efficacy and safety of poractant alfa was evaluated in terms of ventilatory free days during the 21 days after randomization, in adult patients diagnosed with ARDS due to SARS-COV-19 infection.

Each patient randomized to the study treatment received 3 administrations of Curosurf ® with a 24 hours dosing interval. The assessment collection was up to Day 28, when the evaluation occurred at the Intensive Care Unit (ICU), or by phone call if the patient has already been discharged.

Seventy patients were planned to be randomized in the study with a ratio 3:2 (i.e. 42 patients in the poractant alfa arm and 28 in the control arm). The control arm population received Standard of Care (SoC). This study was conducted in United Kingdom (UK), United States of America (US), and Italy.

Overall, 13 patients (Curosurf ® group) and 8 patients (control group) were randomised in the study. Due to low recruitment rate the study was terminated early for non-safety reasons.

Curosurf® is a pulmonary surfactant of natural origin which, when delivered endotracheally (ET). Curosurf® is currently approved for marketing as treatment of premature neonates with RDS or at risk of Respiratory Distress Syndrome (RDS). Chiesi Farmaceutici S.p.A (Chiesi) conducted this study with its porcine-derived surfactant, Curosurf® (poractant alfa), to evaluate the efficacy and safety in ventilated adult patients who were critically unwell in intensive care with SARS-COV-19 ARDS.

ELIGIBILITY:
Inclusion Criteria:

Participants were eligible to be included in the study if the following criteria apply:

1. Male or female ≥18 and ≤ 80 years of age
2. Informed consent for participation in the study (refer to section 15 for detailed inform consent procedure)
3. Positive 2019-nCoV Reverse Transcription Polymerase Chain Reaction (rt-PCR) before randomisation
4. Arterial Partial Pressure of Oxygen/Fraction of Inspired Oxygen (PaO2/FiO2) ratio < 150 mmHg
5. Lung compliance ≤45 ml/cmH20
6. Intubated and artificially ventilated less than 48 hours before the first poractant alfa administration

Exclusion Criteria:

Participants were excluded from the study if any of the following criteria apply:

1. Any contraindications to surfactant administration e.g., pulmonary hemorrhage and pneumothorax)
2. Weight < 40kg
3. Stage 4 severe chronic kidney disease (i.e., Estimated Glomerular Filtration Rate (eGFR) < 30)
4. Pregnancy
5. Administration of any nebulized surfactant in the 48 hours before the first poractant alfa administration
6. Extracorporeal membrane oxygenation (ECMO)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2021-01-06 (Actual); Primary Completion 2022-03-17 (Actual); Study Completion 2022-03-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clark Howard, Prof. /MD, Principal Investigator — University College, London
Locations (6):
- Henry Ford Health System, Detroit, Michigan, United States
- Italy (2):
  - Chiesi site # 14, Bologna
  - Chiesi site #13, Modena
- United Kingdom (3):
  - UCLH and UCL 250 Euston Road, London
  - Chiesi site #4, London
  - Chiesi site # 12, Southampton

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Study Record on EU Clinical Trials Register including results — https://www.clinicaltrialsregister.eu/ctr-search/trial/2020-002632-75/results

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The planned 70 randomised patients in a 3:2 ratio, according to the inclusion and exclusion criteria. This was not achieved; owing to a global improvement in the pandemic situation in the countries where the study was performed (Italy, UK, US), patient recruitment was lower than expected (i.e. 22 patients were randomised, 14 patients and 8 patients in the poractant alfa and control groups, respectively); the study was terminated early before reaching the target sample size.
Groups:
- Control Cohort: Patients receiving standard-of-care (SoC)
- Poractant Alfa Treated Cohort: Patients treated with CUROSURF® (poractant alfa), as an add-on to standard-of-care (SoC)
Period: Overall Study
Arm/Group | Control Cohort | Poractant Alfa Treated Cohort
Started | 8 | 14
Completed | 5 | 9
Not Completed | 3 | 5
Not completed — Death | 2 | 4
Not completed — Lost to Follow-up | 1 | 0
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intention-to-Treat (ITT) population used for this parameter.
Groups:
- Control Cohort: Patients receiving SoC
- Total: Total of all reporting groups
Arm/Group | Control Cohort | Poractant Alfa Treated Cohort | Total
Number analyzed (Participants) | 8 | 13 | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 7 | 12
  >=65 years | 3 | 6 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.0 (18.2) | 63.6 (9.2) | 58.8 (14.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 6 | 10 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 6 | 12 | 18
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Body mass index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 36.44 (9.90) | 29.78 (5.05) | 32.32 (7.78)
Arterial Partial Pressure of Oxygen/Fraction of inspired oxygen (PaO2/FiO2) ratio [Mean (Standard Deviation); unit: Ratio] — The ratio of partial pressure of oxygen in arterial blood (PaO2) to the fraction of inspiratory oxygen concentration (FiO2) is an indicator of pulmonary shunt fraction. PaO2/FiO2 (P/F) ratio is used to classify severity of acute respiratory distress syndrome (ARDS).
  To calculate the P/F Ratio: PaO2 / FIO2. "P" represents PaO2 (arterial pO2) from the arterial blood gas. "F" represents the FIO2 - the fraction (percent) of inspired oxygen that the patient is receiving expressed as a decimal (40% oxygen = FIO2 of 0.40). P divided by F = P/F ratio
  Ratio | 109.70 (51.15) | 111.85 (38.72) | 111.03 (42.62)
Fraction of inspired oxygen (FiO2) [Mean (Standard Deviation); unit: percentage of inspired oxygen] — The fraction of inspired oxygen, FiO2, is an estimation of the oxygen content a person inhales and is thus involved in gas exchange at the alveolar level.
  percentage of inspired oxygen | 70.5 (18.1) | 65.0 (23.2) | 67.1 (21.1)
Sequential Organ Failure Assessment (SOFA) score [Mean (Standard Deviation); unit: score] — Sequential Organ Failure Assessment (SOFA) score is a scoring system that assesses the performance of several organ systems in the body (neurologic, blood, liver, kidney, and blood pressure/hemodynamics) and assigns a score based on the data obtained in each category.
  Total score ranged from 0 to 24 points; to be considered organ failure free, a patient had to have a score of 0.
  score | 7.0 (3.5) | 7.8 (4.6) | 7.5 (4.2)

OUTCOME MEASURES:

1. Primary Outcome: Number of Days Alive and Ventilator-free Days
Description: The number of days alive and ventilator-free days, defined as the number of days the patient is not receiving mechanical ventilation over the 21 days following randomisation.
  Mechanical ventilation was defined as invasive and non-invasive. The patient was defined as free of mechanical ventilation after 12 hours from the suspension of either invasive and non-invasive ventilation. Patients who died or were mechanically ventilated longer than this period were assessed as zero ventilator-free days.
Time Frame: up to 21 days
Population: Intention-to-Treat (ITT) population: all randomised patients who had at least one available evaluation of efficacy after baseline.
  Data was summarised by treatment group using, descriptive statistics.
  Due to low recruitment rate the study was terminated early for non-safety reasons.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Control Cohort | Poractant Alfa Treated Cohort
Number analyzed (Participants) | 8 | 13
days | 4.8 (6.6) | 1.2 (4.2)

2. Secondary Outcome: Percentage of Patients Alive and Free of Respiratory Failure at Day 28
Description: The percentage of patients alive and free of respiratory failure (i.e. without need for mechanical ventilation, extracorporeal membrane oxygenation (ECMO), non-invasive ventilation, or high-flow nasal cannula oxygen delivery) at Day 28.
Time Frame: at Day 28
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Control Cohort | Poractant Alfa Treated Cohort
Number analyzed (Participants) | 8 | 13
percentage of participants | 25.0 | 15.4

3. Secondary Outcome: Number of Days Alive and Ventilator-Free at Day 28
Description: The number of days alive and ventilator-free (i.e. free of any mechanical ventilation for at least 12 hours) at Day 28.
Time Frame: at Day 28
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Control Cohort | Poractant Alfa Treated Cohort
Number analyzed (Participants) | 8 | 13
days | 7.4 (10.2) | 1.7 (6.1)

4. Secondary Outcome: Mortality at Day 21 and Day 28
Description: Mortality at Day 21 and Day 28 of the study by treatment group.
Time Frame: at Day 21 and at Day 28
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Control Cohort | Poractant Alfa Treated Cohort
Number analyzed (Participants) | 8 | 13
Participants
  Dead at Day 21 | 2 | 4
  Dead at Day 28 | 2 | 4

5. Secondary Outcome: Number of Days Alive and Free From Invasive Ventilation at Day 21 and Day 28
Description: The number of days alive and free from invasive ventilation at Day 21 and Day 28 is presented by treatment group.
Time Frame: Day 21 and Day 28
Population: as for outcome 1
Measure: Median (Full Range); unit: days
Arm/Group | Control Cohort | Poractant Alfa Treated Cohort
Number analyzed (Participants) | 8 | 13
days
  Days alive and free from invasive ventilation at Day 21 | 0 [0 to 15] | 0 [0 to 15]
  Days alive and free from invasive ventilation at Day 28 | 0 [0 to 22] | 0 [0 to 22]

6. Secondary Outcome: Number of Days Alive and Free From Non-Invasive Ventilation at Day 21 and Day 28
Description: The number of days alive and free from non-invasive ventilation at Day 21 and Day 28 is presented by treatment group.
Time Frame: Day 21 and Day 28
Population: as for outcome 1
Measure: Median (Full Range); unit: days
Arm/Group | Control Cohort | Poractant Alfa Treated Cohort
Number analyzed (Participants) | 8 | 13
days
  Days alive and free from non-invasive ventilation at Day 21 | 12.5 [0 to 21] | 21.0 [0 to 21]
  Days alive and free from non-invasive ventilation at Day 28 | 19.5 [0 to 28] | 28.0 [0 to 28]

7. Secondary Outcome: Percentage of Patients With Improvement in Severity Status at Day 28 or Discharge (Severity Score: Mild, Moderate, Severe, or Death)
Description: The severity status of patients at baseline and at Day 28/Discharge and the percentage of patients with improvement in severity status (i.e. a decrease of at least 1 point in severity status) at Day 28/Discharge relative to baseline is presented.
  Severity was assessed using a point score system: Severity score was defined as mild, moderate, severe (see below*), or death and was based on PaO2/FiO2 ratio and patient status at Day 28/Discharge and numerically rated from 1-4, respectively. An improvement in severity was defined as a decrease of at least 1 point between baseline and Day 28/Discharge.
  At Day 28 the last follow up evaluation took place on the ICU if, still requiring critical care, or by phone call if the patient has been discharged from ICU by that time.
  *Mild: 200 mmHg < PaO2/FiO2 ratio ≤300 mmHg; Moderate: 100 mmHg < PaO2/FiO2 ratio ≤200 mmHg; Severe: PaO2/FiO2 ratio ≤100 mmHg
Time Frame: Day 28 or Discharge, whichever comes first
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Control Cohort | Poractant Alfa Treated Cohort
Number analyzed (Participants) | 6 | 12
percentage of participants | 50.0 | 25.0

8. Secondary Outcome: Change From Baseline in Arterial Partial Pressure of Oxygen / Fraction of Inspired Oxygen (PaO2/FiO2) Ratio at Each Timepoint
Description: Change from baseline in PaO2/FiO2 ratio measured at each timepoint following administration of each dose in the treatment and control group.
  The change was calculated from two time points as the value at the later time point minus the value at baseline.
  Partial pressure of oxygen (PaO2) is the oxygen pressure in arterial blood. The fraction of inspired oxygen (FiO2) is the concentration of oxygen in the gas mixture.
  The fraction of inspired oxygen (PaO2/FiO2) ratio is widely used in ICUs as an indicator of oxygenation status.
Time Frame: up to 28 days: 6, 12, 24, 30, 36, 48, 54, 60, 72 hours after randomisation, and Day 28
Population: Intention-to-Treat (ITT) population: all randomised patients who had at least one available evaluation of efficacy after baseline.
  Data was summarised by treatment group using, descriptive statistics. Due to low recruitment rate the study was terminated early for non-safety reasons.
  At each time point the number of patients that contributed with a result value is indicated for both study arms.
Measure: Median (Full Range); unit: mmHg
Arm/Group | Control Cohort | Poractant Alfa Treated Cohort
Number analyzed (Participants) | 8 | 13
mmHg
  6 hours | 7.00 [-53.50 to 197.08] | 13.00 [-67.50 to 67.51]
  12 hours: number analyzed (Participants) | 8 | 12
  12 hours | 23.00 [-60.58 to 220.00] | 10.01 [-60.00 to 82.51]
  24 hours | 31.00 [-69.42 to 235.00] | 2.36 [-57.01 to 67.00]
  30 hours: number analyzed (Participants) | 7 | 13
  30 hours | 70.00 [-104.92 to 182.00] | 10.00 [-41.02 to 143.00]
  36 hours | 11.00 [-103.80 to 203.00] | 31.00 [-35.40 to 165.02]
  48 hours | 24.00 [-83.11 to 183.00] | 15.65 [-38.00 to 89.00]
  54 hours: number analyzed (Participants) | 7 | 12
  54 hours | 78.00 [-132.19 to 304.00] | 25.07 [-54.61 to 98.00]
  60 hours: number analyzed (Participants) | 7 | 13
  60 hours | 0.00 [-103.06 to 308.00] | 7.00 [-56.00 to 120.01]
  72 hours: number analyzed (Participants) | 7 | 11
  72 hours | -1.40 [-39.41 to 278.00] | -1.00 [-41.85 to 67.00]
  28 day: number analyzed (Participants) | 2 | 7
  28 day | 53.50 [-21.00 to 128.00] | 20.00 [-93.45 to 135.02]

9. Secondary Outcome: Percentage of Patients Alive and With PaO2/FiO2 Ratio Improvement >20% Compared to Baseline at Each Timepoint
Description: The percentages of patients in categories of PaO2/FiO2 ratio improvement compared to baseline (>20%) at all timepoints post-baseline are summarised by treatment group.
Time Frame: up to 28 days: 6, 12, 24, 30, 36, 48, 54, 60, 72 hours after randomisation and Day 28
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Control Cohort | Poractant Alfa Treated Cohort
Number analyzed (Participants) | 8 | 13
percentage of participants
  6 hours | 37.5 | 46.2
  12 hours: number analyzed (Participants) | 8 | 12
  12 hours | 62.5 | 41.7
  24 hours | 50.0 | 38.5
  30 hours: number analyzed (Participants) | 7 | 13
  30 hours | 57.1 | 38.5
  36 hours | 50.0 | 53.8
  48 hours | 50.0 | 46.2
  54 hours: number analyzed (Participants) | 7 | 12
  54 hours | 71.4 | 58.3
  60 hours: number analyzed (Participants) | 7 | 13
  60 hours | 28.6 | 38.5
  72 hours: number analyzed (Participants) | 7 | 12
  72 hours | 14.3 | 33.3
  28 day: number analyzed (Participants) | 4 | 11
  28 day | 25.0 | 27.3

10. Secondary Outcome: Change From Baseline in Fraction of Inspired Oxygen (FiO2) at Each Timepoint
Description: The FiO2 at baseline and at selected timepoints post-baseline was measured. Results are shown as changes from baseline, summarised by treatment group.
  The change was calculated from two time points as the value at the later time point minus the value at baseline. The unit for the variable is percent (%) and what is reported is an absolute change.
Time Frame: up to 28 days: 6, 12, 24, 30, 36, 48, 54, 60, 72 hours after randomisation and Day 28
Population: as for outcome 1
Measure: Median (Full Range); unit: percent (absolute change)
Arm/Group | Control Cohort | Poractant Alfa Treated Cohort
Number analyzed (Participants) | 8 | 13
percent (absolute change)
  6 hours | -7.2 [-30.0 to 20.0] | 0.0 [-35.0 to 20.0]
  12 hours | -2.5 [-25.0 to 20.0] | -5.0 [-50.0 to 15.0]
  24 hours | 0.0 [-30.0 to 15.0] | 0.0 [-45.0 to 55.0]
  30 hours: number analyzed (Participants) | 7 | 13
  30 hours | -15.0 [-30.0 to 5.7] | -5.0 [-50.0 to 25.0]
  36 hours | -10.0 [-30.0 to 15.0] | -10.0 [-50.0 to 10.0]
  48 hours | -12.5 [-35.0 to 45.7] | 0.0 [-55.0 to 55.0]
  54 hours | -12.5 [-50.0 to 15.7] | -5.0 [-55.0 to 50.0]
  60 hours | 2.5 [-40.0 to 20.0] | -5.0 [-60.0 to 20.0]
  72 hours: number analyzed (Participants) | 8 | 12
  72 hours | -4.9 [-50.0 to 10.0] | 0.0 [-55.0 to 50.0]
  28 day: number analyzed (Participants) | 3 | 8
  28 day | -14.3 [-60.0 to 10.0] | -7.5 [-60.0 to 50.0]

11. Secondary Outcome: Length of ICU Stay (Days) at Day 28
Description: The length of ICU stay (days) at Day 28 is presented by treatment by treatment group. Patients who died or were mechanically ventilated longer than this period were assigned with 28 days.
Time Frame: up to 28 days
Population: as for outcome 1
Measure: Median (Full Range); unit: days
Arm/Group | Control Cohort | Poractant Alfa Treated Cohort
Number analyzed (Participants) | 8 | 13
days | 28.0 [9 to 28] | 28.0 [12 to 28]

12. Secondary Outcome: Percentage of Patients Alive and Out of Intensive Care Unit (ICU) at Day 28
Description: The percentage of patients alive and out of ICU at Day 28 is presented by treatment group.
Time Frame: Day 28
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Control Cohort | Poractant Alfa Treated Cohort
Number analyzed (Participants) | 8 | 13
percentage of participants | 37.5 | 7.7

13. Secondary Outcome: Delta Sequential Organ Failure Assessment (SOFA) Score and Sub-component Measure at Day 3 and Day 28
Description: The Sequential Organ Failure Assessment (SOFA) score is a scoring system that assesses the performance of several organ systems in the body. The SOFA score was used to determine the extent of organ failure at Day 3 and Day 28/Discharge with respect to a pre-randomisation assessment.
  The total score was derived from six sub-scores system categories: respiratory, neurological, cardiovascular, hepatic, coagulation, and renal systems; respective sub-scores were calculated primarily considering PaO2/FiO2 ratio, Glasgow Coma Scale, mean arterial pressure (MAP) or requirement for vasopressor administration, bilirubin levels, platelet levels and creatinine levels or daily urine output.
  A score of 0, 1, 2, 3, or 4) was assigned to each of the six system category. The total score ranged from 0 (min) to 24 (max) points. To be considered organ failure free, a patient had to have a score of 0.
Time Frame: Day 3 and Day 28 or discharge -- whichever comes first
Population: as for outcome 1
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Control Cohort | Poractant Alfa Treated Cohort
Number analyzed (Participants) | 8 | 13
score on a scale
  SOFA score -- Day 3 | 0.5 [-5 to 5] | 0.0 [-5 to 5]
  SOFA score -- Day 28 / Discharge: number analyzed (Participants) | 5 | 8
  SOFA score -- Day 28 / Discharge | -1.0 [-6 to 11] | 0.0 [-4 to 2]
  Respiratory system score -- Day 3 | 0.0 [-1 to 1] | 0.0 [-1 to 1]
  Respiratory system score -- Day 28 / Discharge: number analyzed (Participants) | 5 | 8
  Respiratory system score -- Day 28 / Discharge | -1.0 [-1 to 0] | -0.5 [-1 to 1]
  Neurological system score -- Day 3 | 0.0 [-4 to 2] | 0.0 [0 to 1]
  Neurological system score -- Day 28 / Discharge: number analyzed (Participants) | 5 | 8
  Neurological system score -- Day 28 / Discharge | -2.0 [-4 to 2] | 0.0 [-3 to 0]
  Cardiovascular system score -- Day 3 | 0.0 [-1 to 1] | 0.0 [-3 to 3]
  Cardiovascular system score -- Day 28 / Discharge: number analyzed (Participants) | 5 | 8
  Cardiovascular system score -- Day 28 / Discharge | 0.0 [-1 to 3] | 0.0 [-2 to 1]
  Hepatic system score -- Day 3 | 0.0 [-1 to 0] | 0.0 [-2 to 2]
  Hepatic system score -- Day 28 / Discharge: number analyzed (Participants) | 5 | 8
  Hepatic system score -- Day 28 / Discharge | 0.0 [0 to 1] | 0.0 [0 to 0]
  Coagulatory system score -- Day 3 | 0.0 [-1 to 1] | 0.0 [-1 to 1]
  Coagulatory system score -- Day 28 / Discharge: number analyzed (Participants) | 5 | 8
  Coagulatory system score -- Day 28 / Discharge | 0.0 [-1 to 3] | 0.0 [-1 to 1]
  Renal system score -- Day 3 | 0.0 [0 to 4] | 0.0 [0 to 2]
  Renal system score -- Day 28 / Discharge: number analyzed (Participants) | 5 | 8
  Renal system score -- Day 28 / Discharge | 0.0 [0 to 2] | 0.0 [0 to 0]

14. Secondary Outcome: Percentage of Patients Alive and Free of Organ Failure (SOFA Score=0)
Description: The percentage of patients alive and organ failure free (defined as SOFA score=0) at Day 28/Discharge is presented by treatment group.
  The total score was derived from six sub-scores system categories: respiratory, neurological, cardiovascular, hepatic, coagulation, and renal systems; respective sub-scores were calculated primarily considering PaO2/FiO2 ratio, Glasgow Coma Scale, mean arterial pressure (MAP) or requirement for vasopressor administration, bilirubin levels, platelet levels and creatinine levels or daily urine output.
  A score of 0, 1, 2, 3, or 4) was assigned to each of the six system category. The total score ranged from 0 (min) to 24 (max) points. To be considered organ failure free, a patient had to have a score of 0.
Time Frame: at day 28 or discharge -- whichever comes first
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Control Cohort | Poractant Alfa Treated Cohort
Number analyzed (Participants) | 8 | 13
percentage of participants | 0 | 0

15. Secondary Outcome: Ventilatory Parameter: Tidal Volume -- Change From Baseline in Tidal Volume (mL/kg BW) at All Timepoints up to Day 3 (72 Hours) and at Day 28
Description: Ventilatory parameter: Change from baseline in tidal volume (mL/kg BW) at all timepoints up to Day 3 (72 hours) and at Day 28.
  The change was calculated from two time points as the value at the later time point minus the value at baseline.
  Tidal volume is the amount of air that moves in or out of the lungs with each respiratory cycle.
Time Frame: up to 28 days: 6, 12, 24, 30, 36, 48, 54, 60, 72 hours after randomisation and Day 28
Population: as for outcome 1
Measure: Median (Full Range); unit: mL/kg BW
Arm/Group | Control Cohort | Poractant Alfa Treated Cohort
Number analyzed (Participants) | 8 | 13
mL/kg BW
  6 hours | 1.50 [-101.0 to 152.0] | -1.00 [-90.0 to 93.0]
  12 hours | 4.50 [-67.0 to 194.0] | 13.00 [-170.0 to 129.0]
  24 hours: number analyzed (Participants) | 7 | 13
  24 hours | 15.00 [-252.0 to 166.0] | 0.00 [-170.0 to 147.0]
  30 hours: number analyzed (Participants) | 7 | 13
  30 hours | 61.00 [-53.0 to 514.8] | -18.00 [-119.0 to 79.0]
  36 hours | 54.50 [-219.0 to 532.4] | 13.40 [-67.0 to 146.0]
  48 hours | -34.00 [-125.0 to 512.0] | -17.00 [-160.0 to 230.0]
  54 hours | 7.00 [-250.0 to 521.0] | 30.00 [-116.0 to 320.0]
  60 hours: number analyzed (Participants) | 7 | 13
  60 hours | -8.00 [-129.0 to 233.0] | 17.00 [-141.0 to 256.0]
  72 hours: number analyzed (Participants) | 8 | 12
  72 hours | 73.50 [-272.0 to 271.6] | 11.50 [-136.0 to 234.0]
  28 day: number analyzed (Participants) | 3 | 6
  28 day | 5.00 [-257.0 to 35.8] | -90.50 [-325.0 to -26.0]

16. Secondary Outcome: Ventilatory Parameter: Respiratory Rate -- Change From Baseline in Respiratory Rate (Breaths/Minute) at All Timepoints up to Day 3 (72 Hours) and at Day 28
Description: Ventilatory parameter: Change from baseline in respiratory rate (breaths/minute) at all timepoints up to Day 3 (72 hours) and at Day 28.
  The change was calculated from two time points as the value at the later time point minus the value at baseline.
  Respiratory rate is the number of breaths taken per minute.
Time Frame: up to 28 days: 6, 12, 24, 30, 36, 48, 54, 60, 72 hours after randomisation and Day 28
Population: as for outcome 1
Measure: Median (Full Range); unit: breaths/minute
Arm/Group | Control Cohort | Poractant Alfa Treated Cohort
Number analyzed (Participants) | 8 | 13
breaths/minute
  6 hours | 0.0 [-4.0 to 5.0] | 0.0 [-2.0 to 1.0]
  12 hours | 0.0 [-1.0 to 5.0] | 0.0 [-2.0 to 8.0]
  24 hours | 2.50 [-1.0 to 8.0] | 0.0 [-2.0 to 6.0]
  30 hours: number analyzed (Participants) | 7 | 13
  30 hours | 4.0 [-9.0 to 17.0] | 0.0 [-3.0 to 4.0]
  36 hours | 1.0 [-11.0 to 11.0] | 0.0 [-4.0 to 4.0]
  48 hours | 1.50 [-11.0 to 11.0] | 0.0 [-6.0 to 4.0]
  54 hours | 0.00 [-8.0 to 14.0] | 0.0 [-15.0 to 8.0]
  60 hours | 0.0 [-10.0 to 13.0] | 0.0 [-15.0 to 15.0]
  72 hours: number analyzed (Participants) | 8 | 12
  72 hours | 1.0 [-6.0 to 13.0] | 0.00 [-14.0 to 13.0]
  28 day: number analyzed (Participants) | 3 | 8
  28 day | 10.0 [-6.0 to 12.0] | 14.0 [2.0 to 26.0]

17. Secondary Outcome: Ventilatory Parameter: Dynamic Compliance -- Change From Baseline in Dynamic Compliance (mL/cmH2O) at All Timepoints up to Day 3 (72 Hours) and at Day 28
Description: Ventilatory parameter: Change from baseline in dynamic compliance (mL/cmH2O) at all timepoints up to Day 3 (72 hours) and at Day 28.
  The change was calculated from two time points as the value at the later time point minus the value at baseline.
  Dynamic compliance: is the continuous measurement of pulmonary compliance calculated at each point representing schematic changes during rhythmic breathing. Dynamic compliance monitors both elastic and airway resistance.
Time Frame: up to 28 days: 6, 12, 24, 30, 36, 48, 54, 60, 72 hours after randomisation and Day 28
Population: as for outcome 8
Measure: Median (Full Range); unit: mL/cmH2O
Arm/Group | Control Cohort | Poractant Alfa Treated Cohort
Number analyzed (Participants) | 8 | 13
mL/cmH2O
  6 hours: number analyzed (Participants) | 5 | 12
  6 hours | -1.0 [-4.0 to 9.2] | 0.70 [-6.3 to 13.3]
  12 hours: number analyzed (Participants) | 5 | 13
  12 hours | 0.50 [-4.0 to 15.5] | -0.70 [-4.0 to 3.5]
  24 hours: number analyzed (Participants) | 5 | 11
  24 hours | 1.20 [-11.7 to 6.3] | -0.55 [-5.3 to 2.9]
  30 hours: number analyzed (Participants) | 4 | 12
  30 hours | 7.50 [-1.0 to 46.0] | 1.30 [-0.6 to 188.8]
  36 hours: number analyzed (Participants) | 5 | 12
  36 hours | 3.00 [-1.9 to 63.0] | 2.25 [-0.4 to 6.2]
  48 hours: number analyzed (Participants) | 5 | 12
  48 hours | 2.00 [-10.5 to 103.0] | 0.52 [-12.8 to 14.2]
  54 hours: number analyzed (Participants) | 6 | 12
  54 hours | 1.80 [-23.9 to 105.0] | 0.98 [-4.1 to 11.3]
  60 hours: number analyzed (Participants) | 4 | 12
  60 hours | 0.85 [-5.5 to 7.0] | -0.05 [-3.9 to 5.2]
  72 hours: number analyzed (Participants) | 6 | 11
  72 hours | -1.25 [-25.7 to 7.0] | 0.0 [-10.5 to 14.5]
  28 day: number analyzed (Participants) | 2 | 7
  28 day | -5.25 [-24.5 to 14.0] | -3.10 [-13.0 to 0.7]

18. Secondary Outcome: Ventilatory Parameter: Static Compliance -- Change From Baseline in Static Compliance (mL/cmH2O) at All Timepoints up to Day 3 (72 Hours) and at Day 28
Description: Ventilatory parameter: static compliance -- change from baseline in static compliance (mL/cmH2O) at all timepoints up to Day 3 (72 hours) and at Day 28.
  The change was calculated from two time points as the value at the later time point minus the value at baseline.
  At each time point the number of patients that contributed with a result value is indicated for both study arms.
  Static Compliance: represents pulmonary compliance at a given fixed volume when there is no airflow, and muscles are relaxed.
Time Frame: up to 28 days: 6, 12, 24, 30, 36, 48, 54, 60, 72 hours after randomisation and Day 28
Population: as for outcome 1
Measure: Median (Full Range); unit: mL/cmH2O
Arm/Group | Control Cohort | Poractant Alfa Treated Cohort
Number analyzed (Participants) | 8 | 13
mL/cmH2O
  6 hours: number analyzed (Participants) | 4 | 10
  6 hours | -2.00 [-4.0 to 9.2] | 0.40 [-4.0 to 12.2]
  12 hours: number analyzed (Participants) | 4 | 10
  12 hours | 0.15 [-4.0 to 8.5] | -0.81 [-3.5 to 4.3]
  24 hours: number analyzed (Participants) | 4 | 9
  24 hours | 1.54 [0.0 to 6.3] | -0.40 [-3.6 to 5.1]
  30 hours: number analyzed (Participants) | 3 | 9
  30 hours | 7.00 [-1.0 to 8.0] | 1.30 [0.2 to 12.8]
  36 hours: number analyzed (Participants) | 4 | 9
  36 hours | 2.50 [-1.9 to 7.5] | 2.10 [-0.4 to 6.2]
  48 hours: number analyzed (Participants) | 4 | 9
  48 hours | -3.50 [-10.5 to 7.4] | -0.40 [-5.7 to 9.2]
  54 hours: number analyzed (Participants) | 4 | 8
  54 hours | 1.80 [-23.9 to 7.1] | -0.26 [-3.7 to 6.4]
  60 hours: number analyzed (Participants) | 4 | 9
  60 hours | 0.85 [-5.5 to 7.0] | -0.40 [-3.2 to 5.6]
  72 hours: number analyzed (Participants) | 4 | 8
  72 hours | 3.00 [-25.7 to 7.0] | 0.30 [-1.3 to 13.2]
  28 day: number analyzed (Participants) | 1 | 5
  28 day | -24.50 [-24.5 to -24.5] | -2.70 [-13.0 to 0.7]

19. Secondary Outcome: Ventilatory Parameter: Positive End-Expiratory Pressure (PEEP) -- Change From Baseline in PEEP (cmH2O) at All Timepoints up to Day 3 (72 Hours) and at Day 28
Description: Ventilatory parameter: Positive End-Expiratory Pressure -- Change from baseline in PEEP (cmH2O) at all timepoints up to Day 3 (72 hours) and at Day 28.
  The change was calculated from two time points as the value at the later time point minus the value at baseline.
  At each time point the number of patients that contributed with a result value is indicated for both study arms.
  Positive end-expiratory pressure (PEEP) is the positive pressure that will remain in the airways at the end of the respiratory cycle (end of exhalation) that is greater than the atmospheric pressure in mechanically ventilated patients.
Time Frame: up to 28 days: 6, 12, 24, 30, 36, 48, 54, 60, 72 hours after randomisation and Day 28
Population: as for outcome 1
Measure: Median (Full Range); unit: cmH2O
Arm/Group | Control Cohort | Poractant Alfa Treated Cohort
Number analyzed (Participants) | 8 | 13
cmH2O
  6 hours: number analyzed (Participants) | 8 | 12
  6 hours | 0.00 [-0.3 to 2.0] | 0.00 [-4.0 to 0.1]
  12 hours: number analyzed (Participants) | 8 | 12
  12 hours | 0.50 [0.0 to 2.0] | 0.00 [-2.0 to 0.3]
  24 hours: number analyzed (Participants) | 7 | 12
  24 hours | 2.00 [-3.0 to 2.0] | 0.00 [-4.0 to 7.0]
  30 hours: number analyzed (Participants) | 7 | 12
  30 hours | 0.00 [-4.0 to 2.0] | 0.00 [-4.0 to 1.0]
  36 hours: number analyzed (Participants) | 8 | 12
  36 hours | 0.00 [-5.0 to 5.0] | 0.00 [-4.0 to 1.0]
  48 hours: number analyzed (Participants) | 8 | 12
  48 hours | 0.00 [-8.0 to 3.0] | 0.00 [-4.0 to 1.0]
  54 hours: number analyzed (Participants) | 8 | 12
  54 hours | -0.50 [-10.0 to 3.0] | -0.50 [-7.6 to 1.0]
  60 hours: number analyzed (Participants) | 8 | 12
  60 hours | -0.45 [-10.0 to 3.0] | -0.50 [-6.0 to 1.0]
  72 hours: number analyzed (Participants) | 8 | 11
  72 hours | -1.00 [-10.0 to 3.0] | 0.00 [-2.0 to 1.0]
  28 day: number analyzed (Participants) | 3 | 7
  28 day | -3.20 [-11.8 to -1.0] | -2.00 [-4.0 to 0.2]

20. Secondary Outcome: Ventilatory Parameter: Peak Inspiratory Pressure -- Change From Baseline in Peak Inspiratory Pressure (cmH2O) at All Timepoints up to Day 3 (72 Hours) and at Day 28
Description: Ventilatory parameter: Peak Inspiratory Pressure -- Change from baseline in peak inspiratory pressure (cmH2O) at all timepoints up to Day 3 (72 hours) and at Day 28.
  The change was calculated from two time points as the value at the later time point minus the value at baseline.
  At each time point the number of patients that contributed with a result value is indicated for both study arms.
  Peak inspiratory pressure (PIP) is the highest level of pressure applied to the lungs during inhalation. In mechanical ventilation the number reflects a positive pressure in centimetres of water pressure (cmH2O).
Time Frame: up to 28 days: 6, 12, 24, 30, 36, 48, 54, 60, 72 hours after randomisation and Day 28
Population: as for outcome 1
Measure: Median (Full Range); unit: cmH2O
Arm/Group | Control Cohort | Poractant Alfa Treated Cohort
Number analyzed (Participants) | 8 | 13
cmH2O
  6 hours: number analyzed (Participants) | 8 | 12
  6 hours | 0.00 [-18.0 to 5.0] | 0.00 [-8.0 to 4.0]
  12 hours | 2.00 [-0.1 to 5.0] | 0.00 [-8.0 to 3.4]
  24 hours: number analyzed (Participants) | 7 | 12
  24 hours | 3.00 [-4.1 to 6.0] | -0.50 [-8.0 to 2.2]
  30 hours: number analyzed (Participants) | 6 | 13
  30 hours | 1.00 [-4.7 to 6.0] | -2.00 [-6.0 to 5.0]
  36 hours: number analyzed (Participants) | 7 | 13
  36 hours | 3.00 [-4.7 to 6.0] | -1.00 [-8.0 to 2.1]
  48 hours | 0.00 [-5.4 to 10.0] | -2.00 [-8.0 to 8.0]
  54 hours | 2.00 [-5.5 to 8.0] | -3.00 [-8.0 to 1.0]
  60 hours: number analyzed (Participants) | 7 | 13
  60 hours | 0.00 [-6.1 to 7.0] | -3.00 [-7.0 to 2.0]
  72 hours: number analyzed (Participants) | 8 | 12
  72 hours | 4.50 [-7.0 to 12.0] | -3.00 [-13.0 to 4.0]
  28 day: number analyzed (Participants) | 3 | 7
  28 day | 4.00 [-3.5 to 5.0] | -4.00 [-16.0 to 8.0]

21. Secondary Outcome: Ventilatory Parameter: Plateau Pressure -- Change From Baseline in Plateau Pressure (cmH2O) at All Timepoints up to Day 3 (72 Hours) and at Day 28
Description: Ventilatory parameter: Plateau Pressure -- Change from baseline in plateau pressure (cmH2O) at all timepoints up to Day 3 (72 hours) and at Day 28.
  The change was calculated from two time points as the value at the later time point minus the value at baseline.
  At each time point the number of patients that contributed with a result value is indicated for both study arms.
  Plateau pressure is the pressure that is applied by the mechanical ventilator to the small airways and alveoli.
Time Frame: up to 28 days: 6, 12, 24, 30, 36, 48, 54, 60, 72 hours after randomisation, and Day 28
Population: as for outcome 1
Measure: Median (Full Range); unit: cmH2O
Arm/Group | Control Cohort | Poractant Alfa Treated Cohort
Number analyzed (Participants) | 8 | 13
cmH2O
  6 hours: number analyzed (Participants) | 4 | 9
  6 hours | 1.25 [0.0 to 3.0] | -1.00 [-8.0 to 2.0]
  12 hours: number analyzed (Participants) | 4 | 10
  12 hours | 2.00 [0.0 to 3.0] | -1.50 [-8.0 to 2.0]
  24 hours: number analyzed (Participants) | 6 | 10
  24 hours | 0.50 [-5.0 to 6.0] | -1.50 [-8.0 to 2.0]
  30 hours: number analyzed (Participants) | 4 | 9
  30 hours | 0.00 [-1.0 to 6.0] | -3.00 [-7.0 to 1.0]
  36 hours: number analyzed (Participants) | 5 | 10
  36 hours | 1.00 [-2.0 to 4.0] | -2.00 [-8.0 to 1.0]
  48 hours: number analyzed (Participants) | 5 | 9
  48 hours | 3.00 [-4.0 to 10.0] | -3.00 [-8.0 to 1.0]
  54 hours: number analyzed (Participants) | 6 | 10
  54 hours | 1.50 [-4.0 to 10.0] | -3.50 [-8.0 to 1.0]
  60 hours: number analyzed (Participants) | 6 | 10
  60 hours | 0.50 [-5.0 to 7.0] | -2.50 [-7.0 to 2.0]
  72 hours: number analyzed (Participants) | 6 | 9
  72 hours | 1.50 [-8.0 to 11.0] | -3.00 [-8.0 to 3.0]
  28 day: number analyzed (Participants) | 2 | 5
  28 day | 2.00 [-2.0 to 6.0] | -4.00 [-16.0 to 15.7]

22. Secondary Outcome: Blood Gas Analysis Acid-base Balance Parameters: Change From Baseline in Blood Gas Analysis Acid-base Balance Parameters -- pH
Description: Change from baseline in blood gas analysis acid-base balance parameters -- pH.
  The change was calculated from two time points as the value at the later time point minus the value at baseline.
  Arterial blood gas was measured at 6, 12, 24, 30, 36, 48, 54, 60 and 72 hours after randomisation and up to Day 28 or till the patient was discharged from the ICU - whichever occurred earlier.
Time Frame: up to 28 days: 6, 12, 24, 30, 36, 48, 54, 60, 72 hours after randomisation, and Day 28
Population: as for outcome 1
Measure: Median (Full Range); unit: pH
Arm/Group | Control Cohort | Poractant Alfa Treated Cohort
Number analyzed (Participants) | 8 | 13
pH
  6 hours: number analyzed (Participants) | 8 | 12
  6 hours | 0.0000 [-0.020 to 0.100] | 0.0080 [-0.240 to 0.127]
  12 hours | 0.0050 [-0.080 to 0.080] | 0.0100 [-0.150 to 0.149]
  24 hours | 0.0315 [-0.110 to 0.150] | 0.0160 [-0.150 to 0.110]
  30 hours: number analyzed (Participants) | 7 | 13
  30 hours | 0.0300 [-0.090 to 0.150] | 0.0100 [-0.120 to 0.210]
  36 hours | 0.0050 [-0.110 to 0.180] | 0.0260 [-0.080 to 0.170]
  48 hours | 0.0050 [-0.100 to 0.160] | 0.0300 [-0.320 to 0.170]
  54 hours: number analyzed (Participants) | 7 | 12
  54 hours | 0.0500 [-0.150 to 0.457] | 0.0185 [-0.230 to 0.170]
  60 hours: number analyzed (Participants) | 7 | 13
  60 hours | -0.0500 [-0.140 to 0.348] | 0.0000 [-0.369 to 0.140]
  72 hours: number analyzed (Participants) | 7 | 11
  72 hours | 0.0400 [-0.170 to 0.270] | 0.0120 [-0.369 to 0.180]
  28 day: number analyzed (Participants) | 3 | 8
  28 day | -0.0400 [-0.050 to -0.021] | 0.0500 [-0.010 to 0.230]
  ICU Discharge: number analyzed (Participants) | 0 | 1
  ICU Discharge |  | 0.0450 [0.045 to 0.045]

23. Secondary Outcome: Change From Baseline in Blood Gas Analysis Acid-base Balance Parameter -- Partial Pressure of Carbon Dioxide (pCO2)
Description: Change from baseline in blood gas analysis acid-base balance parameter -- pCO2.
  The change was calculated from two time points as the value at the later time point minus the value at baseline.
  Arterial blood gas was measured at 6, 12, 24, 30, 36, 48, 54, 60 and 72 hours after randomisation and up to Day 28 or till the patient was discharged from the ICU - whichever occurred earlier.
Time Frame: up to 28 days: 6, 12, 24, 30, 36, 48, 54, 60, 72 hours after randomisation, and Day 28
Population: as for outcome 1
Measure: Median (Full Range); unit: mmHg
Arm/Group | Control Cohort | Poractant Alfa Treated Cohort
Number analyzed (Participants) | 8 | 13
mmHg
  6 hours: number analyzed (Participants) | 8 | 12
  6 hours | -2.210 [-10.40 to 5.00] | 1.535 [-14.25 to 49.00]
  12 hours | -0.150 [-11.00 to 11.00] | 1.730 [-21.76 to 22.10]
  24 hours | -2.610 [-19.00 to 18.00] | -2.000 [-29.26 to 18.10]
  30 hours: number analyzed (Participants) | 7 | 13
  30 hours | -5.700 [-11.40 to 10.60] | 1.880 [-21.50 to 20.25]
  36 hours | -3.350 [-15.00 to 23.00] | 1.720 [-13.50 to 12.00]
  48 hours | 2.500 [-11.00 to 10.20] | 0.300 [-14.50 to 16.00]
  54 hours: number analyzed (Participants) | 7 | 11
  54 hours | -0.600 [-38.50 to 13.60] | -1.500 [-13.00 to 30.00]
  60 hours: number analyzed (Participants) | 7 | 13
  60 hours | 3.400 [-5.40 to 28.00] | -0.230 [-10.00 to 19.00]
  72 hours: number analyzed (Participants) | 7 | 11
  72 hours | 0.000 [-10.87 to 33.00] | 0.750 [-18.00 to 33.10]
  28 day: number analyzed (Participants) | 3 | 7
  28 day | 6.150 [-8.00 to 52.00] | 12.000 [-13.40 to 30.01]
  ICU Discharge: number analyzed (Participants) | 0 | 1
  ICU Discharge |  | -9.600 [-9.60 to -9.60]

24. Secondary Outcome: Change From Baseline in Blood Gas Analysis Acid-base Balance Parameter -- Partial Pressure of Oxygen (pO2)
Description: Change from baseline in blood gas analysis acid-base balance parameter -- pO2.
  The change was calculated from two time points as the value at the later time point minus the value at baseline.
  Arterial blood gas was measured at 6, 12, 24, 30, 36, 48, 54, 60 and 72 hours after randomisation and up to Day 28 or till the patient was discharged from the ICU - whichever occurred earlier.
Time Frame: up to 28 days: 6, 12, 24, 30, 36, 48, 54, 60, 72 hours after randomisation, and Day 28
Population: as for outcome 1
Measure: Median (Full Range); unit: mmHg
Arm/Group | Control Cohort | Poractant Alfa Treated Cohort
Number analyzed (Participants) | 8 | 13
mmHg
  6 hours: number analyzed (Participants) | 8 | 12
  6 hours | 0.500 [-9.00 to 210.01] | 6.550 [-14.60 to 165.61]
  12 hours | 12.500 [-8.85 to 158.70] | 1.000 [-20.78 to 50.85]
  24 hours | 7.000 [-6.30 to 82.70] | 1.100 [-19.28 to 98.26]
  30 hours: number analyzed (Participants) | 7 | 13
  30 hours | 3.000 [-11.40 to 181.10] | 2.000 [-25.28 to 29.10]
  36 hours | 7.000 [-13.30 to 171.10] | 2.600 [-16.35 to 28.35]
  48 hours | 6.250 [-10.30 to 63.10] | 0.000 [-19.20 to 52.00]
  54 hours: number analyzed (Participants) | 7 | 11
  54 hours | 4.300 [-23.33 to 116.10] | 2.250 [-29.56 to 43.00]
  60 hours: number analyzed (Participants) | 7 | 13
  60 hours | 15.000 [-13.05 to 156.10] | 0.000 [-32.26 to 21.00]
  72 hours: number analyzed (Participants) | 7 | 11
  72 hours | 6.000 [-6.30 to 103.10] | 5.100 [-7.00 to 50.25]
  28 day: number analyzed (Participants) | 3 | 7
  28 day | 8.100 [-7.00 to 33.00] | -7.700 [-26.78 to 34.50]
  ICU Discharge: number analyzed (Participants) | 0 | 1
  ICU Discharge |  | -10.730 [-10.73 to -10.73]

25. Secondary Outcome: Change From Baseline in Blood Gas Analysis Acid-base Balance Parameter -- Bicarbonate (HCO3)
Description: Change from baseline in blood gas analysis acid-base balance parameter -- Bicarbonate (HCO3).
  The change was calculated from two time points as the value at the later time point minus the value at baseline.
  Measured at 6-12-24h after each poractant alfa administration up to 72 hours and at similar timepoints in the control group (6, 12, 24, 30, 36, 48, 54, 60 and 72 hours after randomisation) and then every 24 hours till the patient is discharged from the ICU
Time Frame: up to 28 days: 6, 12, 24, 30, 36, 48, 54, 60, 72 hours after randomisation, and Day 28
Population: as for outcome 1
Measure: Median (Full Range); unit: mmol/L
Arm/Group | Control Cohort | Poractant Alfa Treated Cohort
Number analyzed (Participants) | 8 | 13
mmol/L
  6 hours: number analyzed (Participants) | 8 | 12
  6 hours | 1.05 [-1.1 to 19.3] | 0.70 [-3.8 to 4.4]
  12 hours | 1.10 [-0.6 to 5.0] | 1.30 [-2.4 to 5.6]
  24 hours | 1.65 [-3.5 to 6.7] | 1.80 [-2.4 to 5.5]
  30 hours: number analyzed (Participants) | 7 | 13
  30 hours | 2.30 [-3.0 to 5.7] | 2.30 [-2.4 to 6.3]
  36 hours | 1.75 [-2.8 to 7.5] | 2.70 [-2.7 to 6.9]
  48 hours | 1.60 [-4.1 to 7.8] | 3.50 [-13.4 to 7.7]
  54 hours: number analyzed (Participants) | 7 | 11
  54 hours | 0.80 [-19.1 to 8.9] | 2.10 [-11.4 to 5.8]
  60 hours: number analyzed (Participants) | 7 | 13
  60 hours | 3.30 [-3.9 to 10.7] | 2.80 [-2.9 to 9.1]
  72 hours: number analyzed (Participants) | 7 | 11
  72 hours | 3.00 [-4.5 to 10.4] | 4.00 [0.6 to 11.6]
  28 day: number analyzed (Participants) | 3 | 7
  28 day | 1.90 [-6.4 to 33.0] | 13.20 [5.3 to 17.5]
  ICU Discharge: number analyzed (Participants) | 0 | 1
  ICU Discharge |  | -3.90 [-3.90 to -3.90]

26. Secondary Outcome: Change From Baseline in Blood Parameter -- Lactate
Description: Change from baseline in blood parameter -- Lactate
  The change was calculated from two time points as the value at the later time point minus the value at baseline.
  At each time point the number of patients that contributed with a result value is indicated for both study arms.
  Arterial blood lactate was measured at 6, 12, 24, 30, 36, 48, 54, 60, and 72 hours after randomisation and up to Day 28 or till the patient was discharged from the ICU - whichever occurred earlier.
Time Frame: up to 28 days: 6, 12, 24, 30, 36, 48, 54, 60, 72 hours after randomisation, and Day 28
Population: as for outcome 1
Measure: Median (Full Range); unit: mmol/L
Arm/Group | Control Cohort | Poractant Alfa Treated Cohort
Number analyzed (Participants) | 8 | 13
mmol/L
  6 hours: number analyzed (Participants) | 6 | 12
  6 hours | 0.05 [-0.5 to 1.1] | -0.05 [-1.0 to 0.5]
  12 hours: number analyzed (Participants) | 6 | 13
  12 hours | 0.55 [-0.8 to 1.8] | 0.20 [-1.1 to 0.6]
  24 hours: number analyzed (Participants) | 7 | 13
  24 hours | -0.10 [-0.4 to 1.3] | -0.10 [-0.9 to 0.5]
  30 hours: number analyzed (Participants) | 6 | 13
  30 hours | 0.30 [-0.4 to 1.2] | 0.00 [-0.8 to 1.0]
  36 hours: number analyzed (Participants) | 6 | 13
  36 hours | 0.55 [-0.8 to 1.5] | -0.10 [-0.9 to 9.8]
  48 hours: number analyzed (Participants) | 6 | 13
  48 hours | -0.10 [-0.7 to 1.5] | -0.10 [-1.2 to 17.6]
  54 hours: number analyzed (Participants) | 6 | 11
  54 hours | 0.25 [-0.3 to 1.3] | 0.00 [-1.5 to 21.6]
  60 hours: number analyzed (Participants) | 7 | 13
  60 hours | 0.10 [-1.0 to 1.4] | -0.10 [-1.8 to 19.6]
  72 hours: number analyzed (Participants) | 7 | 11
  72 hours | -0.20 [-1.3 to 0.9] | -0.10 [-1.1 to 1.0]
  28 day: number analyzed (Participants) | 3 | 7
  28 day | -0.60 [-1.0 to 1.4] | -0.10 [-1.2 to 0.4]
  ICU Discharge: number analyzed (Participants) | 0 | 1
  ICU Discharge |  | -2.30 [-2.30 to -2.30]

27. Secondary Outcome: Mortality -- TEAEs Leading to Death
Description: The incidence of treatment-emergent adverse event (TEAEs) leading to death is presented by treatment group.
Time Frame: up to day 28
Population: Safety Population: all randomised patients (who received at least one dose of the study treatment if poractant alfa-treated).
Measure: Count of Participants; unit: Participants
Arm/Group | Control Cohort | Poractant Alfa Treated Cohort
Number analyzed (Participants) | 8 | 13
Participants | 2 | 3

ADVERSE EVENTS:
Time Frame: From screening procedures (Day 0) to the end of the study (Day 28).
Description: Analysis of adverse events (AEs) was performed on TEAEs, defined as AEs that started at or after treatment start (for the poractant alfa group) or at or after randomisation (for the control group).
  Safety set (SAF) was used to evaluate AEs and serious AEs (SAEs). The SAF included all enrolled patients, except for one, who was randomised to receive poractant alfa was not treated. All patients included in the SAF were also included in the ITT.
Arm/Group | Control Cohort | Poractant Alfa Treated Cohort
All-Cause Mortality (participants affected / at risk) | 2/8 | 4/13
Serious Adverse Events (participants affected / at risk) | 3/8 | 5/13
Other Adverse Events (participants affected / at risk) | 5/8 | 11/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Cohort (N=8) | Poractant Alfa Treated Cohort (N=13)
Atrioventricular block (Cardiac disorders) | 0 (0) | 1 (1)
Cardiogenic shock (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Right ventricular failure (Cardiac disorders) | 1 (1) | 1 (1)
Bicytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pneumatosis intestinalis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 0 (0)
Nosocomial infection (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Soft tissue injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Cerebral artery embolism (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral disorder (Nervous system disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Cohort (N=8) | Poractant Alfa Treated Cohort (N=13)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Impaired gastric emptying (Gastrointestinal disorders) | 1 (1) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hyperpyrexia (General disorders) | 1 (1) | 0 (0)
Hyperthermia (General disorders) | 0 (0) | 1 (1)
Haemophagocytic lymphohistiocytosis (Immune system disorders) | 1 (1) | 0 (0)
Aspergillus infection (Infections and infestations) | 0 (0) | 1 (1)
Bacterial sepsis (Infections and infestations) | 0 (0) | 1 (1)
Empyema (Infections and infestations) | 1 (1) | 0 (0)
Enterococcal infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumococcal infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 2 (3) | 2 (3)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 2 (2)
Pneumonia klebsiella (Infections and infestations) | 0 (0) | 1 (1)
Proteus infection (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 2 (2)
Septic shock (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal infection (Infections and infestations) | 1 (1) | 1 (1)
Urinary tract infection bacterial (Infections and infestations) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Refractoriness to platelet transfusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (1)
Neutrophil count increased (Investigations) | 0 (0) | 1 (1)
Transaminases increased (Investigations) | 1 (1) | 0 (0)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
Hypertension (Vascular disorders) | 1 (1) | 1 (1)

LIMITATIONS AND CAVEATS:
Once the impact of the Covid 19 pandemic significantly declined and intubated patients with acute respiratory distress syndrome (ARDS) outcome became rare, the Sponsor considered it unfeasible to maintain efforts to recruit further patients into the study. Thus, due to low recruitment, the study was terminated early for non-safety reasons.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Chiesi can publish and/or present any results of this study at scientific meetings, and to submit the clinical trial data to national and international Regulatory Authorities. Chiesi reserves the right to use such data for industrial purposes. Investigators will inform Chiesi before using the results of the study for publication or presentation, and agree to provide the Sponsor with a copy of the proposed presentation. Data from individual study sites must not be published separately.

DOCUMENTS (2):
  • Study Protocol (2021-03-02): https://cdn.clinicaltrials.gov/large-docs/33/NCT04502433/Prot_000.pdf
  • Statistical Analysis Plan (2022-07-27): https://cdn.clinicaltrials.gov/large-docs/33/NCT04502433/SAP_001.pdf